CLINICAL TRIAL: NCT02351310
Title: Effects of Antenatal Corticosteroids in Patients With Early (22 - 23w6d) Threatened Preterm Birth
Brief Title: Effectiveness of ACS in Extreme Preemies
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decided not to pursue this study.
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBX0031
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Preterm Labor; Premature Birth
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Betamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Betamethasone (Active Comparator): Betamethasone: 12 mg given intramuscularly (IM), 24 hours apart or if as in some hospitals occasionally occurs and betamethasone is unavailable - • 4 doses of Dexamethasone IM 6 mg, 12 hours apart
  Interventions: Drug: Betamethasone
- Normal Saline (Placebo Comparator): Quantity Sufficient (QS) of Normal Saline (NS) given intramuscularly (IM), 24 hours apart or if hospital is using Dexamethasone in place of Betamethasone then administer NS x 4 doses 12 hours apart
  Interventions: Genetic: Placebo

INTERVENTIONS:
Drug: Betamethasone — Course of ACS given intramuscularly (2 doses of 12 mg, 24 hours apart)
  Other Names: ACS
  Arms: Betamethasone
Genetic: Placebo — Course of placebo drug given intramuscularly (2 doses of normal saline (of equal quantity) 24 hours apart).
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
This is a randomized prospective clinical study that will evaluate the effects of antenatal corticosteroid administration (ACS) vs. placebo in singleton pregnancies who are threatening to deliver prematurely between 22 0/7 and 23 6/7 weeks on admission with the goal of improving composite neonatal mortality and morbidity.

DETAILED DESCRIPTION:
The purpose of this study to evaluate the effects of antenatal corticosteroid administration (ACS) vs. placebo in patients who are threatening to deliver prematurely with well-established gestational ages between 22 0/7 and 23 6/7 weeks at the time of admission. If the delivery can be safely delayed at least 3 hours and there is no contraindication to steroid administration, the patient is eligible to be randomized. Randomization will be blinded to the patient and the staff caring for the patient and will be stratified by gestational age: those at 22 0/7 to 22 6/7 weeks and those at 23 0/7 weeks to 23 6/7 weeks. Randomized patients will be assignment to either active drug or placebo at the doses and frequencies below:

* 2 doses of Betamethasone, 12 mg intramuscularly (IM), 24 hours apart, or if as in some hospitals occasionally occurs and betamethasone is unavailable -
* 4 doses of Dexamethasone IM 6 mg, 12 hours apart.

Remainder of care will be at the discretion of the clinician.

Randomized 22 0/7 - 22 6/7:

For patients randomized between 22 0/7 and 22 6/7 weeks and who are undelivered > 24 0/7 weeks, the decision as to whether to administer an additional course or courses of ACS will also be at the discretion of the clinician.

Randomized 23 0/7 to 23 6/7:

For those patients randomized at 23 0/7 to 23 6/7 weeks and who remain undelivered > 24 0/7 weeks and < 1 week after study medication was administered, a second blinded set of medications/placebos will be provided. For patients who received Betamethasone (or dexamethasone) placebo will be provided and for those who received placebo Betamethasone will be provided.(for both at the doses described in 3.4.3). In this group, at any time > 24 0/7 weeks and less than one week of the previous dose, if the clinician feels the patient is still at risk for delivering, this second blinded set of study drugs will be administered. This will allow the patient to receive at least one actual course of ACS if undelivered at 24w0d. In this group, if the patient remains undelivered at > 25 weeks, administration of an open label course of ACS will be at the discretion of the MD.

Primary Outcome of this study is composite morbidity and mortality. The N on this study is 68 (34 in each group)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at time of study entry
* Gestational age between 22 0/7 to 23 6/7 weeks, inclusive at time of randomization regardless of whether the provider and patient decide to consider the fetus viable and provide obstetric interventions and cesarean section if needed.
* Singleton pregnancy
* Threatening to deliver by the best estimate of the clinician within the ensuing week
* Thought by the clinician to be able to delay delivery at least 3 hours from the time of randomization.
* Desired Pregnancy
* All clinical complications related to or leading to delivery except those listed as exclusion criteria are eligible. All of the following clinical complications are eligible including but not limited to:

  * premature labor,
  * incompetent cervix with or without prolapsing membranes,
  * Preterm Premature Rupture of the membranes (PPROM),
  * chorioamnionitis,
  * all hypertensive disorders of pregnancy,
  * vaginal bleeding due to placenta previa, abruption or unknown etiology,
  * being delivered for medical complication of pregnancy, and others.

Exclusion Criteria:

* Maternal history of insulin dependent diabetes
* Known congenital fetal anomaly
* Known Hydrops fetalis with this current pregnancy
* Severe intrauterine growth restriction < 10% percentile
* Patient receiving corticosteroids for other maternal indications other than for fetal lung maturity
* Patient with h/o HIV or active Tuberculosis.
* Any other known contraindication to corticosteroids

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Composite Neonatal Morbidity | First 30 days after birth
  Defined as one or more of the following: fetal death, neonatal death within 30 days of delivery, respiratory distress syndrome (oxygen requirement, clinical diagnosis and consistent chest x-ray), bronchopulmonary dysplasia (requirement for oxygen support at 30 days of life), severe intraventricular hemorrhage (IVH) (grades III or IV), periventricular leukomalacia, blood culture proven sepsis, necrotizing enterocolitis (NEC).

SECONDARY OUTCOMES:
Preterm Birth prior to 34weeks gestational age. | From entry into the study until 34 weeks gestational age.
  Preterm birth that occurs between the time of enrollment into the study (22w0d-23w6d) until 34w6d.
Respiratory Distress Syndrome (RDS) | First 30 days after birth
  RDS is defined as compatible symptoms with radiographically confirmed hyaline membrane disease or ￼ with respiratory insufficiency of prematurity requiring ventilator support are present.
Birth Weight | Measured at time of birth
  newborns birth weight
Newborn Head Circumference measurement | Measured at time of birth
  Measurement of newborn head circumference done at time of birth.
Need for Newborn Surfactant Therapy | First 30 days after birth
  administration of newborn surfactant therapy within the first 30day of life.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Garite, MD, Study Director — Pediatrix

IPD SHARING:
Plan to Share IPD: No